CLINICAL TRIAL: NCT06812650
Title: Effects of Diaphragmatic Breathing and Relaxation Exercises in Patients With Gastroesophageal Reflux
Brief Title: Breathing Exercises in Patients With Gastroesophageal Reflux
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Tarik Ozmen, Professor, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBU-FTR-2024/1814
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-02

CONDITIONS: Reflux Disease, Gastro-Esophageal
Keywords: Breathing Exercises; Relaxation; Quality of Life; Anxiety
MeSH Terms: conditions — Gastroesophageal Reflux; Anxiety Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medical Treatment (Active Comparator)
  Interventions: Other: Medical treatment
- Exercise (Experimental): The exercise program will consist of diaphragmatic breathing exercises and progressive muscle relaxation exercises.
  Interventions: Other: Medical treatment; Other: Exercise

INTERVENTIONS:
Other: Medical treatment — Patients will continue their routine medical treatment for gastroesophageal reflux disease.
Other: Exercise — The exercise program will consist of diaphragmatic breathing exercises and progressive muscle relaxation exercises. Diaphragmatic breathing exercises will be performed for 8 weeks, 5 days a week, twice a day, for 15 minutes each time.
  Arms: Exercise

SUMMARY:
The aim of this study was to examine the effects of diaphragmatic breathing exercises combined with relaxation exercises on patient-reported reflux symptoms, quality of life, anxiety, and depression levels in patients diagnosed with gastroesophageal reflux.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease is a pathological condition in which various symptoms and/or complications occur as a result of the escape of stomach contents into the esophagus, oral cavity, or lungs. Gastroesophageal reflux disease is largely associated with various respiratory diseases such as chronic cough, idiopathic pulmonary fibrosis, chronic obstructive pulmonary disease, and asthma. Accordingly, respiratory function deterioration may be observed in spirometric measurements. Increased symptom burden in gastroesophageal reflux patients has been associated with poor quality of life, sleep disturbances, and decreased physical function and productivity. However, increased anxiety and depression levels in patients are also closely related to reflux symptoms.At the esophagogastric junction, the lower esophageal sphincter and the surrounding crura of the diaphragm constitute an important part of the protective mechanism against reflux. The crural diaphragm, which contracts during inspiration, acts as an additional external sphincter. Since the crural diaphragm is a striated muscle structure, it is possible to improve its function with exercise. Eherer et al. (2012) examined the effects of diaphragmatic breathing exercises performed for 30 minutes per day for 4 weeks on pH levels, quality of life, and medication use in patients with non-erosive reflux. As a result of the study, they found that quality of life increased and acid exposure decreased.The recurrence rate and maintenance treatment requirement after treatment are high in reflux patients. Proton pump inhibitor drugs commonly used in treatment may have various side effects in the long term. Although the diaphragm muscle is an important part of the protective mechanism against reflux, there are few studies investigating the effects of applications targeting this muscle on reflux.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who do not have cardiopulmonary, mental, connective tissue, metabolic, or other diseases that may prevent exercise
* Individuals who do not have body mass index >35 or <18
* Individuals who are not addicted to alcohol or cigarettes
* Individuals who are between the ages of 18 and 65
* Individuals who are diagnosed with non-erosive reflux will be included in the study.

Exclusion Criteria:

* Individuals with a history of gastrointestinal surgery
* Individuals who are pregnant or breastfeeding
* Individuals who have hiatal hernia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Gastroesophageal Reflux Disease Questionnaire | Eight weeks
  Reflux symptoms will be assessed with the Gastroesophageal Reflux Disease Questionnaire. The frequency of 6 questions regarding heartburn, regurgitation, dyspepsia, nausea, need for medication, and sleep disturbances in the last 7 days are scored. The total score can range from 0-18.
Gastroesophageal Reflux Disease- Quality of Life | Eight weeks
  The scale aims to measure how regurgitation and pyrosis symptoms have affected the patient's daily life in the last 7 days. It consists of 16 questions under 4 main headings: daily activity, treatment effect, diet and psychological well-being. It is evaluated with a five-point Likert-type scale. A low total score indicates that the quality of life has also decreased.

SECONDARY OUTCOMES:
The Hospital Anxiety and Depression Scale | Eight weeks
  The Hospital Anxiety and Depression Scale will be used to assess anxiety and depression. HADS was developed to assess anxiety disorders and depression in patients in hospital clinics other than psychiatry. Each question in the scale, consisting of a total of 14 questions, is evaluated between 0 and 3 points. Increasing scores represent higher levels of anxiety and depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Private Maras Health Services, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No